CLINICAL TRIAL: NCT04084496
Title: A Phase II Study With mFOLFIRINOX as Adjuvent Chemotherapy for Resectable Pancreas Carcinoma
Brief Title: mFOLFIRINOX as Adjuvent Chemotherapy in Treating Chinese Pancreatic Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mFOLFIRINOX_PC
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; adjuvant chemotherapy; FOLFIRINOX
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOLFIRINOX (Experimental): Patients will receive mFOLFIRINOX every 2 weeks: Oxaliplatin 65 mg/m2 IV over 3 hours on Day 1; Irinotecan 150 mg/m2 IV over 90 minutes on Day 1; Leucovorin(l-LV) 200 mg/m2 IV over 2 hours on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion.
  Interventions: Drug: Folfirinox

INTERVENTIONS:
Drug: Folfirinox — Patients will receive mFOLFIRINOX every 2 weeks: Oxaliplatin 65 mg/m2 IV over 3 hours on Day 1; Irinotecan 150 mg/m2 IV over 90 minutes on Day 1; Leucovorin(l-LV) 200 mg/m2 IV over 2 hours on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion.

SUMMARY:
Although FOLFIRINOX regimen was recently presented to be effective as adjuvant chemotherapy for resectable pancreatic cancer in selected patients who have good physical condition, there is still insufficient evidence on this regimen in treating resectable pancreatic cancer patients in China. Since for many tumors, different races may show different responses to the same regimen, we design this open phase Ⅱ study to evaluate the the efficacy and safety of mFOLFIRINOX as adjuvant chemotherapy for resectable pancreatic cancer in China.

DETAILED DESCRIPTION:
This is a phase II study. Patients with resectable pancreatic carcinoma will receive adjuvant chemotherapy of FOLFIRINOX for 6 months.

Primary endpoint is the disease free survival. Secondary endpoints are overall survival, safety and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas without distant metastases.
* Receive radical resection of pancreatic cancer
* No prior cytostatic chemotherapy
* Female and male patients > 18 and <=79 years using contraception
* ECOG ≤ 1
* Patient has adequate bone marrow and organ function
* Absolute Neutrophil Count (ANC) ≥ 2.0 x 109/L Platelets ≥ 90 x 109/L Hemoglobin ≥ 90 g/L
* Patient has adequate liver function AST and ALT not more than 2.5 times ULN (not more than 5.0 times ULN if there is liver metastasis) Serum bilirubin ≤ 1.2 x ULN Creatinine ≤ 1.25 times ULN
* Good compliance
* Written informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Distant metastasis.
* Patients with severe gastrointestinal hemorrhage which need frequent blood transfusions.
* Refuse to take appropriate contraceptive measures (including male patients).
* Allergic to Oxaliplatin, Irinotecan, Leucovorin or 5-Fluorouracil.
* Severe systemic disease out of control such as unstable or uncompensated respiratory, cardiac, liver, renal diseases.
* Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment, (with the exception of non-melanoma skin cancer or cervical carcinoma in situ).
* Psychiatric illness that would prevent the patient from giving informed consent.
* Patient is concurrently using other antineoplastic agent
* Patient has used investigational antineoplastic agent within 4 weeks prior to entry.
* Known HIV-positivity.
* No history of chronic diarrhea, nausea or vomit.
* No ≥ grade 2 sensory peripheral neuropathy.
* A history of transmural myocardial infarction (within 6 months prior to entry), congestive heart failure, and unstable angina.
* Infectious disease or inflammation with body temperature ≥ 38 ℃.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | up to 24 months
  From the date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Overall survival | up to 24 months
  From the date of first drug administration until the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Li, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided